CLINICAL TRIAL: NCT04231968
Title: A Randomized, Double-blind, Placebo-controlled, 2-part Study of Orally Administered AK0529 to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics and Antiviral Effect of Multiple Doses in Hospitalized Infants With Respiratory Syncytial Virus Infection
Brief Title: A Study of AK0529 in Chinese Infants Hospitalized With RSV
Acronym: AIRFLO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK0529-2003
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — ziresovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK0529 (Experimental): Participants who are randomized to the experimental arm will receive AK0529 twice daily for five days .
  Interventions: Drug: AK0529
- Placebo (Placebo Comparator): Participants in the control arm will be administered placebo at the matching dosage levels of active medications.
  Interventions: Drug: Matching placebo of AK0529

INTERVENTIONS:
Drug: AK0529 — AK0529 capsule will be orally administered at the twice-daily dosing levels of 10 mg, 20 mg, or 40 mg for five days based on the patient's weight.
  Other Names: ziresovir
  Arms: AK0529
Drug: Matching placebo of AK0529 — The placebo capsule was made with the same smell and appearance as AK0529 but without the active ingredients and will be orally administered per the same treatment schedule as those in the experimental arm.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, phase III study to be conducted in infants hospitalized with RSV infection in China. The main objectives of this study are to investigate the efficacy and safety of AK0529 in Chinese infants.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female patients of any ethnicity with an age-adjusted for any prematurity of ≥1 month and ≤24 months.
* Diagnosis of RSV infection by any virological means within 36 hours preceding the initial dose.
* The time from the onset caused by RSV infection to the first dose should be ≤ 7 days. Time of onset is defined as the time the first respiratory or systemic signs or symptoms of RSV infection confirmed by the investigator.
* Body weight ≥ 2.5 kg and ≤ 20 kg at screening.
* For patients aged <12 months, an occipitofrontal head circumference should be within the normal range for age and gender.
* Bronchiolitis score ≥ 5.
* The parent/legal guardian must have provided written informed consent for the patient to participate.

Main Exclusion Criteria:

* Patients who have used any prohibited medications within 72 hours prior to expected administration and those who have used inhaled or systemic glucocorticosteroids within 24 hours prior to administration.
* Patients (or mothers of patients younger than 6 months of age) with a known HIV-positive history or patients highly suspected HIV-positive by the investigator.
* Patients with known co-infection with influenza virus.
* Patient known to have pneumonia caused by bacterial infection.
* Patients requiring vasopressors or vasoactive drugs at the time of enrollment.
* Concurrent gastrointestinal conditions that could seriously, in the opinion of the investigator, prejudice absorption of the Investigational Medicinal Product.
* Bronchopulmonary dysplasia requiring assisted ventilation at the time of enrolment, except for the result of RSV infection.
* Patients at risk for hypercapnia based on their medical history, except for the result of RSV infection.
* Patient with airway malformations and congenital heart diseases, except for isolated patent ductus arteriosus and/or patent foramen ovale.
* Renal failure including renal abnormalities likely to be associated with renal insufficiency.
* Clinical evidence of hepatic decompensation.
* Symptomatic because of congenital metabolic abnormality.
* Chronic or persistent feeding difficulties.
* Known or suspected to have primary immunodeficiency disease.
* Any active or uncontrolled respiratory, cardiac, hepatic, central nervous system or renal disease unrelated to RSV infection at baseline, or any other medical condition that in the opinion of the investigator renders the patient unsuitable for enrolment; in case of any question, discuss such cases with the sponsor's medical monitor.
* A history of epilepsy or seizures including febrile seizures.
* History of family history of high allergies or allergies to multiple substances, or presence of severe rash that in the opinion or the investigator renders the patient unsuitable for enrollment.
* The patient's parent or guardian is an employee of the investigator or the study site with direct involvement in the proposed study or other studies under the direction of that investigator of the study site, or any family members of the employees or the investigator.
* Participation in an investigational drug or device study within 30 days prior to the date of screening.
* Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 311 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Clinically significant change from baseline in bronchiolitis score on Day 3 | From Baseline (Pre-dose on Day 1) to Day 3 (48 hours)
  To demonstrate that AK0529 is superior to placebo in terms of changes from baseline in bronchiolitis signs and symptoms score.
  The differences of change in the bronchiolitis score are to be evaluated between the AK0529 and placebo arms after treatment. The total score is reported with a range from 0 to 12. Generally, each score component has a range of values from 0 to 3. A decreasing value of the total score represents a clinical improvement. Unless otherwise noted, the last non-missing measurement/assessment before the first dose of the investigational product is defined as the Baseline measurement. If a measurement/evaluation is performed on the same day of the first dose of the investigational product, these measurements will be considered as Baselines.

SECONDARY OUTCOMES:
Change from baseline in RSV (Respiratory syncytial virus) VL(viral load ) on Day 5 | From Baseline (Pre-dose on Day 1) to Day 5 (96 hours)
  To evaluate the antiviral effects of AK0529. The antiviral effects in infants hospitalized with RSV are to be determined by measuring the differences in viral load determined by RT-PCR between the AK0529 and placebo arms after treatment.
Proportions of subjects with a reduction from baseline in clinical bronchiolitis score ≥ 2 after treatment | From Baseline (Pre-dose on Day 1) to Day 14
Proportions of subjects with a reduction from baseline in clinical bronchiolitis score ≥ 3 after treatment | From Baseline (Pre-dose on Day 1) to Day 14
Proportions of subjects with a reduction from baseline in clinical bronchiolitis score ≥ 4 after treatment | From Baseline (Pre-dose on Day 1) to Day 14
Proportions of subjects with a reduction from baseline in clinical bronchiolitis score ≥ 5 after treatment | From Baseline (Pre-dose on Day 1) to Day 14
Proportions of subjects with symptom remission on Day 3 after treatment | Day 3 (48 hours)
  Symptom remission is defined as a reduction in clinical bronchiolitis score to 1 or 0 after treatment.
Proportions of subjects with symptom remission at other visits after treatment | From Baseline (Pre-dose on Day 1) to Day 14 (except for Day 3)
  Symptom remission is defined as a reduction in clinical bronchiolitis score to 1 or 0 after treatment.
Proportions of subjects with ≥ 75% reduction from baseline in bronchiolitis score on Day 3 after treatment | Day 3 (48 hours)
Proportions of subjects with ≥ 75% reduction from baseline in bronchiolitis score at other visits after treatment | From Baseline (Pre-dose on Day 1) to Day 14 (except for Day 3)
Proportions of subjects with disease remission on Day 3 after treatment | From Baseline (Pre-dose on Day 1) to Day 3 (48 hours)
  Disease remission is defined as a reduction in bronchiolitis score to 1 or 0 after treatment, without non-invasive positive pressure ventilation or assisted mechanical ventilation or supplemental oxygen therapy.
Proportions of subjects with disease remission at other visits after treatment. | From Baseline (Pre-dose on Day 1) to Day 14 (except for Day 3)
  Disease remission is defined as a reduction in bronchiolitis score to 1 or 0 after treatment, without non-invasive positive pressure ventilation or assisted mechanical ventilation or supplemental oxygen therapy.
Time from the first dose to symptom remission | From Baseline (Pre-dose on Day 1) to Day 14
  Symptom remission is defined as a reduction in clinical bronchiolitis score to 1 or 0 after treatment.
Time from the first dose to a zero general symptom score for subjects with general symptoms sub-scores equal to 3 at baseline | From Baseline (Pre-dose on Day 1) to Day 14
  The General Symptom score is part of the Bronchiolitis Score and has only two scores, 3 and 0. A normal patient is a 0, and the presence of irritable, lethargic, poor feeding is rated as 3.
Time from the first dose to a ≥ 75% reduction in bronchiolitis score | From Baseline (Pre-dose on Day 1) to Day 14
Time from the first dose to disease remission | From Baseline (Pre-dose on Day 1) to Day 14
  Disease remission is defined as a reduction in bronchiolitis score to 1 or 0 after treatment, without non-invasive positive pressure ventilation or assisted mechanical ventilation or supplemental oxygen therapy.
Change in bronchiolitis score and percentage change from baseline at each visit after treatment (except Day 3) | From Baseline (Pre-dose on Day 1) to Day 14 (except Day 3)
Change from baseline in bronchiolitis sub-score at each visit after treatment | From Baseline (Pre-dose on Day 1) to Day 14
Proportions of subjects with the change in bronchiolitis sub-score values at each visit after treatment | From Baseline (Pre-dose on Day 1) to Day 14
Proportions of subjects achieving a ≥ 50% reduction from baseline in bronchiolitis score after treatment | From Baseline (Pre-dose on Day 1) to Day 14
Proportions of subjects achieving a ≥ 90% reduction from baseline in bronchiolitis score after treatment | From Baseline (Pre-dose on Day 1) to Day 14
Respiratory sequelae of subjects from the end of the safety observation period to Month 6 | From Day 14 to Month 6
  The assessment of respiratory sequelae involves evaluating the frequency, duration, and treatment related to wheezing recurrences and the presence of confirmed asthma.
Respiratory sequelae of subjects from the end of the safety observation period to the end of the second year | From Day 14 to end of Year 2
  The assessment of respiratory sequelae involves evaluating the frequency, duration, and treatment related to wheezing recurrences and the presence of confirmed asthma.
Analysis of subjects admitted to intensive care unit (ICU) for diseases related to RSV infection | From Baseline to the end of ICU
  Analyzed by the number of admissions, duration of admission, and the duration from the first dose to the end of ICU.
Analysis of subjects receiving non-invasive positive pressure ventilation or assisted mechanical ventilation | From Baseline to Day 14
  Analyzed by the number of subjects receiving non-invasive positive pressure ventilation or assisted mechanical ventilation, duration of such ventilation, and the time from the first dose to the end of assisted ventilation.
Analysis of subjects receiving supplemental oxygen therapy | From first treatment to Day 14
  Analyzed by the number of subjects receiving supplemental oxygen therapy, duration of such therapy, and the time from the first dose to supplemental oxygen therapy.
Proportions of subjects with RSV VL below the lower limit of quantification (LLOQ) on Day 5 after treatment | Day 5 (96hours)
Proportions of subjects with RSV VL below the LLOQ at other visits | From Baseline (Pre-dose on Day 1) to Day 14 (except Day 5)
Change from baseline in RSV VL at each visit except Day 5 after treatment | From Baseline (Pre-dose on Day 1) to Day 14 (except Day 5)
Area under the curve of RSV VL from baseline to the last measurement | From Baseline (Pre-dose on Day 1) to Day 14
Analysis of clinical efficacy of AK0529 in different subgroups | From Baseline to Day 14
  Analyzed in different subgroups categorized by, at a minimum, months of age, severity of baseline Bronchiolitis Score, time from onset of RSV infection to first dose, RSV viral subtypes, baseline RSV VL classifications, and doses.
Proportion of subjects with adverse events (AEs) occurring during the study | From Baseline to Day 14
  To evaluate the safety and tolerability of AK0529.
Proportion of subjects with serious adverse events (SAEs) occurring during the study | From Baseline to Day 14
  To evaluate the safety and tolerability of AK0529.
Proportion of subjects who withdraw from the study due to AEs during the study | From Baseline to Day 14
  To evaluate the safety and tolerability of AK0529.
Maximum plasma concentration of AK0529 (Cmax) | At 3 and 24 hours after the first dose and on Day 6 (120 hours)
  PK parameters of AK0529 and its metabolites using population pharmacokinetic (POP-PK) and other appropriate methods.
Plasma drug trough concentration of AK0529 (Ctrough) | At 3 and 24 hours after the first dose and on Day 6 (120 hours)
  PK parameters of AK0529 and its metabolites using population pharmacokinetic (POP-PK) and other appropriate methods.
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) | At 3 and 24 hours after the first dose and on Day 6 (120 hours)
  PK parameters of AK0529 and its metabolites using population pharmacokinetic (POP-PK) and other appropriate methods.
Apparent total body clearance (CL/F) | At 3 and 24 hours after the first dose and on Day 6 (120 hours)
  PK parameters of AK0529 and its metabolites using population pharmacokinetic (POP-PK) and other appropriate methods.
Apparent volume of distribution (Vz/F) | At 3 and 24 hours after the first dose and on Day 6 (120 hours)
  PK parameters of AK0529 and its metabolites using population pharmacokinetic (POP-PK) and other appropriate methods.
Elimination half-life (t½) | At 3 and 24 hours after the first dose and on Day 6 (120 hours)
  PK parameters of AK0529 and its metabolites using population pharmacokinetic (POP-PK) and other appropriate methods.

OTHER OUTCOMES:
RSV VL and primary and selected secondary efficacy measurements | From Baseline to Day 14
  To evaluate the relationship of antiviral effects of AK0529 to the primary and key secondary efficacy measurements.
Selective primary efficacy, secondary efficacy, and safety measures for the pharmacokinetic-pharmacodynamic (PK-PD) analysis | From Baseline to Day 6
  To evaluate the PK-PD correlation between PK parameters and the values of bronchiolitis score and VL, including their respective changes.
Proportions of subjects with mutations at 20 reported sites associated with RSV fusion inhibitor-resistant mutations in RSV F genesequences after treatment compared to baseline | From Baseline to Day 14
  To sequence the F gene of RSV in nasopharyngeal samples to the monitoring on the development of AK0529 resistance mutation. RSV F gene sequencing was performed with nasopharyngeal samples of subjects using Sanger sequencing.
Proportions of subjects detected with other respiratory disease-associated viruses at baseline | Baseline (Pre-dose on Day 1)
  To detect other common respiratory viruses in nasopharyngeal samples. Detection of respiratory disease-associated viruses includes coronaviruses, adenoviruses, metapneumoviruses, rhinoviruses, enteroviruses, influenza A viruses, influenza B viruses, parainfluenza viruses, and other viruses in baseline nasopharyngeal samples from subjects using microfluidic microarray methods.
Changes in respiratory rate during the study | From Baseline through Day 6
  To explore the difference in respiratory rate (bpm) with clinical significance between subjects on AK0529 and those on placebo.
Changes in heart rate during the study | From Baseline through Day 6
  To explore the difference in heart rate/pulse (bpm) with clinical significance between subjects on AK0529 and those on placebo.
Changes in body temperature during the study | From Baseline through Day 6
  To explore the difference in body temperature (Celsius) with clinical significance between subjects on AK0529 and those on placebo.
Changes in systolic blood pressure during the study | From Baseline through Day 6
  To explore the difference in systolic blood pressure (mmHg) with clinical significance between subjects on AK0529 and those on placebo.
Changes in diastolic blood pressure during the study | From Baseline through Day 6
  To explore the difference in diastolic blood pressure (mmHg) with clinical significance between subjects on AK0529 and those on placebo.
Changes in SpO2 during the study | From Baseline through Day 6
  To explore the difference in SpO2 (%) with clinical significance between subjects on AK0529 and those on placebo.
Duration of hospitalization of subjects with RSV infection | From the day of patient admission to the day of patient discharge
  To explore the differences in other clinical measurements between subjects on AK0529 and those on placebo.
Time from first dose to discharge of subjects with RSV infection | From Baseline (Day 1) to the day of patient discharge
  To explore the differences in other clinical measurements between subjects on AK0529 and those on placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chen, MD, Study Director — yu.chen@arkbiosciences.com
Locations (28):
- China (28):
  - Beijing Children's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Hunan Provincial People's Hospital, Changsha
  - West China Women's and Children's Hospital, Chengdu
  - Children's Hospital of Chongqing Medical University, Chongqing
  - Guangzhou Women and Children's Medical Center, Guangzhou
  - The Children's Hospital of Zhejiang University School of Medicine, Hangzhou
  - Liaocheng People's Hospital, Liaocheng
  - Jiangxi Provincial Children's Hospital, Nanchang
  - Children's Hospital of Nanjing Medical University, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanjing
  - Hainan Third People's Hospital, Sanya
  - Children's Hospital of Shanghai, Shanghai
  - Shanghai Children's Medical Center, Shanghai
  - Shengjing Hospital of China Medical University, Shengyang
  - Shenzhen Children's Hospital, Shenzhen
  - Children's Hospital of Soochow University, Suzhou
  - Tianjin Children's Hospital, Tianjin
  - The Second Affiliated Hospital and Yuying Children's Hospital of WMU, Wenzhou
  - Wuhan Children's Hospital, Wuhan
  - Wuxi Children's Hospital, Wuxi
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xiamen Maternity and Child Healthcare Hospital, Xiamen
  - Henan Children's Hospital, Zhengzhou
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Boai Hospital of Zhongshan, Zhongshan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Zhao W, Zhang X, Zhang L, Guo R, Huang H, Lin L, Liu F, Chen H, Shen F, Wu J, Huang X, Zhu X, Li F, Zou G, Chien J, Humphries M, Lu Q, Wu JZ, Zhao S, Liu H, Ni X; AIRFLO Study Group. Efficacy and safety of ziresovir in hospitalised infants aged 6 months or younger with respiratory syncytial virus infection in China: findings from a phase 3 randomised trial with 24-month follow-up. Lancet Child Adolesc Health. 2025 May;9(5):325-336. doi: 10.1016/S2352-4642(25)00067-7. PMID 40246359
- [Derived] Zhao S, Shang Y, Yin Y, Zou Y, Xu Y, Zhong L, Zhang H, Zhang H, Zhao D, Shen T, Huang D, Chen Q, Yang Q, Yang Y, Dong X, Li L, Chen Z, Liu E, Deng L, Jiang W, Cheng H, Nong G, Wang X, Chen Y, Ding R, Zhou W, Zheng Y, Shen Z, Lu X, Hao C, Zhu X, Jia T, Wu Y, Zou G, Rito K, Wu JZ, Liu H, Ni X; AIRFLO Study Group. Ziresovir in Hospitalized Infants with Respiratory Syncytial Virus Infection. N Engl J Med. 2024 Sep 26;391(12):1096-1107. doi: 10.1056/NEJMoa2313551. PMID 39321361